CLINICAL TRIAL: NCT06348147
Title: An Attenuated Schedule Dara-RVd Induction for Patients With Newly Diagnosed Multiple Myeloma Who Are Eligible for Autologous Stem Cell Transplantation
Brief Title: Dara-RVd Induction for Newly Diagnosed Multiple Myeloma With Autologous Stem Cell Transplantation
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: budget
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC2323
Record Dates: First submitted 2024-03-28; First posted 2024-04-04 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Newly Diagnosed Multiple Myeloma; Multiple Myeloma; Autologous Stem Cell Transplantation
Keywords: Daratumumab; lenalidomide; bortezomib; dexamethasone
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Lenalidomide; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Daratumumab, lenalidomide, bortezomib, and dexamethasone (Experimental): Subjects with newly diagnosed multiple myeloma (NDMM) are eligible for standard-of-care autologous stem cell transplantation (ASCT) and receive daratumumab, lenalidomide, bortezomib, and dexamethasone (Dara-RVd).
  Interventions: Biological: Daratumumab; Drug: Lenalidomide; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Biological: Daratumumab — Daratumumab is a CD38-directed cytolytic antibody indicated for the treatment of adults with multiple myeloma. 1800 mg will be given subcutaneously according to its standard package insert schedule.
Drug: Lenalidomide — Lenalidomide will be administered, once daily orally on Days 1-21 of a 28-day
Drug: Bortezomib — Bortezomib is a proteasome inhibitor indicated for the treatment of adult patients with multiple myeloma, will be given subcutaneously once weekly on days 1, 8, and 15 of every 28 day cycle.
Drug: Dexamethasone — Dexamethasone is a glucocorticoid.

SUMMARY:
This Phase II hybrid decentralized trial will examine the effect of daratumumab-based quadruplet induction therapy administered at an attenuated schedule in subjects with newly diagnosed multiple myeloma (NDMM) who are eligible for standard-of-care autologous stem cell transplantation (ASCT). Daratumumab, lenalidomide, bortezomib, and dexamethasone (Dara-RVd) have recently become a standard induction regimen for patients with NDMM who are eligible for ASCT in the United States. As implemented in clinical trials, Dara-RVd involves twice weekly bortezomib administration, which is inconvenient for patients and may result in increased rates of limiting toxicity, such as peripheral neuropathy. Adoption of alternate schedules involving once-weekly bortezomib is common in real-world practice, however a paucity of prospective data supporting this practice exists.

This study examines the efficacy of an attenuated Dara-RVd schedule involving once-weekly bortezomib dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent was obtained to participate in the study and HIPAA authorization for release of personal health information. Subjects are willing and able to comply with study procedures based on the judgment of the investigator.
2. Age ≥18 years at the time of consent.
3. Eastern Cooperative Oncology Group (ECOG) ≤ 2
4. Subjects with Multiple Myeloma.

Exclusion Criteria:

1. Active infection requiring systemic therapy or other serious infection within 14 days prior to study treatment.
2. Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
The rate of achievement of bone marrow minimal residual disease (MRD) negativity | At completion of stem cell transplantation (60 days)
  The rate of achievement of bone marrow minimal residual disease (MRD) negativity will be defined as the percentage of subjects achieving MRD negativity as determined by next-generation flow cytometry.

SECONDARY OUTCOMES:
Progression Free Survival (PFS ) | Up to 2 years
  PFS will be defined as the time from the start of study treatment until progression per revised Uniform Response Criteria by the International Myeloma Working Group (IMWG) or death from any cause.
  Complete response (CR): Negative immunofixation of serum and urine, the disappearance of soft tissue plasmacytomas, and <5% plasma cells in bone marrow (BM). Stringent complete response (sCR): CR plus normal free light chains (FLC) ratio and absence of clonal plasma cells in BM biopsy. Very good partial response (VGPR):-Serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M component plus urine M component <100/24h. Partial response (PR) ≥50% reduction of serum M-protein & reduction in 24-hour (24h) urinary M-protein by ≥90% or to <200 mg/24h and if present at baseline, a ≥ 50% reduction in the size soft tissue plasmacytomas.
Stringent complete response (sCR) | At completion of stem cell transplantation (60 days)
  Stringent complete response (sCR) will be defined according to the standard International Myeloma Working Group (IMWG) response criteria for multiple myeloma.
  Complete response (CR): Negative immunofixation of serum and urine, the disappearance of soft tissue plasmacytomas, and <5% plasma cells in bone marrow (BM). Stringent complete response (sCR): CR plus normal free light chains (FLC) ratio and absence of clonal plasma cells in BM biopsy. Very good partial response (VGPR):-Serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M component plus urine M component <100/24h. Partial response (PR) ≥50% reduction of serum M-protein & reduction in 24-hour (24h) urinary M-protein by ≥90% or to <200 mg/24h and if present at baseline, a ≥ 50% reduction in the size soft tissue plasmacytomas.
Overall Survival (OS) | Up to 2 years
  OS will be defined as the time from the start of treatment to death from any cause.
Therapeutic discontinuation | Up to 2 years
  Therapeutic discontinuation will be defined as a treatment discontinuation of all drugs for any reason.
Time to first response | Up to 2 years
  Time to first response will be defined as time from the start of study treatment until the first achievement of at least a partial response (PR) by IMWG criteria or better.
  Complete response (CR): Negative immunofixation of serum and urine, the disappearance of soft tissue plasmacytomas, and <5% plasma cells in bone marrow (BM). Stringent complete response (sCR): CR plus normal free light chains (FLC) ratio and absence of clonal plasma cells in BM biopsy. Very good partial response (VGPR):-Serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M component plus urine M component <100/24h. Partial response (PR) ≥50% reduction of serum M-protein & reduction in 24-hour (24h) urinary M-protein by ≥90% or to <200 mg/24h and if present at baseline, a ≥ 50% reduction in the size soft tissue plasmacytomas.
Time to best response | Up to 2 years
  The time to best response will be defined as the time from the start of study treatment until the time at which a patient's best response according to IMWG criteria is achieved.
  Complete response (CR): Negative immunofixation of serum and urine, the disappearance of soft tissue plasmacytomas, and <5% plasma cells in bone marrow (BM). Stringent complete response (sCR): CR plus normal free light chains (FLC) ratio and absence of clonal plasma cells in BM biopsy. Very good partial response (VGPR):-Serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M component plus urine M component <100/24h. Partial response (PR) ≥50% reduction of serum M-protein & reduction in 24-hour (24h) urinary M-protein by ≥90% or to <200 mg/24h and if present at baseline, a ≥ 50% reduction in the size soft tissue plasmacytomas.
Maximum depth of response (from PR to CR, including sCR) | Up to 2 years
  The maximum depth of response (from PR to CR, including sCR) will be determined based on IMWG criteria.
  Complete response (CR): Negative immunofixation of serum and urine, the disappearance of soft tissue plasmacytomas, and <5% plasma cells in bone marrow (BM). Stringent complete response (sCR): CR plus normal free light chains (FLC) ratio and absence of clonal plasma cells in BM biopsy. Very good partial response (VGPR):-Serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M component plus urine M component <100/24h. Partial response (PR) ≥50% reduction of serum M-protein & reduction in 24-hour (24h) urinary M-protein by ≥90% or to <200 mg/24h and if present at baseline, a ≥ 50% reduction in the size soft tissue plasmacytomas.
Overall response rate (ORR) | Up to 2 years
  ORR will be defined as the percentage of subjects achieving a partial response (PR) or better according to IMWG criteria.
  Complete response (CR): Negative immunofixation of serum and urine, the disappearance of soft tissue plasmacytomas, and <5% plasma cells in bone marrow (BM). Stringent complete response (sCR): CR plus normal free light chains (FLC) ratio and absence of clonal plasma cells in BM biopsy. Very good partial response (VGPR):-Serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M component plus urine M component <100/24h. Partial response (PR) ≥50% reduction of serum M-protein & reduction in 24-hour (24h) urinary M-protein by ≥90% or to <200 mg/24h and if present at baseline, a ≥ 50% reduction in the size soft tissue plasmacytomas.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel M Rubinstein, MD, MSCI, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials